CLINICAL TRIAL: NCT07312760
Title: Existential Distress in Advanced Cancer: Pragmatic Randomized Controlled Trial of a Short-term Psychodynamic Psychotherapy (ORPHYS) Compared to Treatment as Usual (TAU)
Brief Title: Existential Distress in Advanced Cancer: Comparing a Short-term Psychodynamic Psychotherapy (ORPHYS) to Treatment as Usual (TAU)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: University Düsseldorf (Other); Wuerzburg University Hospital (Other); University of Kassel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DKH70116803
Record Dates: First submitted 2025-12-05; First posted 2025-12-31 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Advanced Cancer, Various, NOS
Keywords: Advanced cancer; Psycho-Oncology; Psychodynamic Psychotherapy; Demoralization; End-of-life; Randomized Controlled Trial; Existential Distress; Psychological Intervention
MeSH Terms: conditions — Pyloric Stenosis, Hypertrophic; Death | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Model Description
Who Masked: Investigator, Outcomes Assessor
Masking Description: Masking Description
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ORPHYS (ShORt term psychodynamic psychotherapy adapted to serious PHYSical illness) (Experimental)
  Interventions: Behavioral: ORPHYS (ShORt-term psychodynamic psychotherapy in serious PHYSical illness)
- TAU (Treatment As Usual: standard psycho-oncological care) (Active Comparator)
  Interventions: Behavioral: TAU (Treatment As Usual: Standard psycho-oncological care)

INTERVENTIONS:
Behavioral: ORPHYS (ShORt-term psychodynamic psychotherapy in serious PHYSical illness) — ORPHYS is a manualized individual psychotherapy that was specifically designed for patients with serious physical illness (Philipp et al., 2024). Patients receive 15-31 weekly therapy sessions of 50 minutes length. ORPHYS takes into account the individual meaning of illness in the context of internalized motives and fears. ORPHYS aims to help patients gain consciousness of related existential conflict. The treatment supports reflection on current relational experiences in the context of realistic, illness-related fears. Identifying patients' dysfunctional relationship patterns, which represent patients' unconscious fantasies about the responsiveness and availability of others and making them accessible to the patient during therapy is expected to increase mentalization and, thus, emotional flexibility to balance extreme affective states. Emotional containment and supportive interventions are the basis for ORPHYS.
  Arms: ORPHYS (ShORt term psychodynamic psychotherapy adapted to serious PHYSical illness)
Behavioral: TAU (Treatment As Usual: Standard psycho-oncological care) — Patients receive routine psycho-oncological care as provided by the study centers. TAU includes individual sessions provided by physicians or master-level psychologists with experience in psycho-oncological care. There is no restriction on the minimum or maximum number of sessions.
  Arms: TAU (Treatment As Usual: standard psycho-oncological care)

SUMMARY:
The psychological challenges faced by patients with incurable cancer and their caregivers include an uncertain future, fear of dying and uncontrollable suffering, grief, and loneliness. In a significant subgroup, this challenge is associated with significant fear and existential distress. This distress can manifest itself, for example, in the form of demoralization, a state of despair and hopelessness in which the possibilities for coping seem exhausted. Although open discussions about fears at the end of life are becoming increasingly important, little is known about how patients with high existential distress can best be supported to promote quality of life.

The aim of the study is to test the effectiveness of the newly developed individual psychotherapy ORPHYS (ShORt-term psychodynamic psychotherapy in serious PHYSical illness) in reducing existential distress. To this end, a randomly selected half of the participants who receive ORPHYS treatment will be compared with a second group who receive the standard routine psycho-oncological treatment TAU (Treatment As Usual). The level of distress caused by demoralization will be used for the comparison. A total of 160 patients with advanced cancer will be included in the study.

Due to improved treatment options, life expectancy for advanced cancer has increased significantly. This means that patients and their families must deal with the existential tension between uncertainty and a focus on life. The treatment is intended to contribute to providing the best possible support for patients who suffer from uncertainty and fears at the end of life.

DETAILED DESCRIPTION:
Background: As improvements in systemic anti-cancer treatments have extended survival, patients with advanced cancer and their family caregivers face the existential tension between engaging in life and coping with uncertainty about illness trajectory and course of treatment. For a subgroup, this tension is associated with overwhelming fear and existential distress. Existential distress is often characterized by demoralization, a state of despair and hopelessness in which coping skills are exhausted and patients are unable to see something positive in the future. Such adjustment difficulties may increase the risk of poor quality of life and suicidality, as well as impair prognostic awareness and patient-clinician communication. Despite growing interest in open conversations about end-of-life issues, little is known about how clinicians can best support patients experiencing high levels of existential distress in order to facilitate psychological adaptation at the end of life.

Objective: To evaluate the effectiveness of ORPHYS (ShORt-term psychodynamic psychotherapy in serious PHYSical illness) in a pragmatic randomized controlled trial. The intervention group receives 15-31 sessions of ORPHYS, a manualized individual psychotherapy that flexibly integrates uncovering and holding treatment elements. The control group receives usual psycho-oncological care (TAU). The primary outcome is demoralization as assessed by the Demoralization Scale-II. Secondary outcomes include diagnosis of affective, anxiety and stress-related disorders, death anxiety, dignity-related distress, and quality of life.

Methods: The investigators will conduct a two-arm parallel randomized controlled trial with an active control group. Patients will be assessed pre-intervention and after 3, 6, 9, and 12 months. The target sample size is 160 participants before randomization. The investigators will recruit patients with stage III/IV solid tumors or advanced hematological cancer and clinically significant existential distress from psycho-oncology clinics and referring oncologists at Hamburg, Düsseldorf, and Würzburg Comprehensive Cancer Centers. Outcome assessments will be conducted via diagnostic interviews and self-report questionnaires. Linear mixed models will examine outcome differences between trial arms. A confirmatory test of the group contrast at 6 months-follow-up will be conducted.

Discussion: Due to an aging population and prolonged survival, there is a growing demand to help patients deal with existential challenges. The study will contribute to knowledge about how clinicians can best help patients with advanced cancer who substantially struggle with uncertainty at the end of life.

ELIGIBILITY:
Inclusion Criteria:

* UICC stage III/IV solid tumor or advanced hematological cancer
* Physical condition at beginning of treatment sufficient for outpatient treatment
* Existential distress due to at least one of the following concerns: loss of hope, demoralization, fear of the future, loneliness, death anxiety, sense of isolation, death wishes
* Severity of distress: significant subjective distress and impairment in functioning

Exclusion Criteria:

* Acute suicidality with concrete or impending intent to follow through (suicide plan)
* diagnosis of a substance dependence, substance abuse, or psychotic disorder (exception: tobacco-related disorders)
* Inability to adhere to a psychotherapeutic setting
* Other current psychotherapeutic or psycho-oncological treatment according to TAU definition
* Insufficient German to give informed consent and complete self-report questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Demoralization assessed via the Demoralization Scale-II (DS-II; Robinson et al., 2016; Koranyi et al., 2021) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 3-point Likert scale from 0 (never) to 2 (often), with a total score ranging from 0 to 32. Higher scores indicate higher demoralization.

SECONDARY OUTCOMES:
Diagnosis of affective disorders, anxiety disorders, trauma- and stressor-related disorders assessed via Diagnostic and Statistical Manual of Mental Disorders-5 (SCID-5; Beesdo-Baum, 2019) | Day 0, Month 6, Month 12
  Presence of the following mental disorders is indicated with "yes" or "no" based on SCID-5 criteria: Major depression, Persistent depressive disorder, Bipolar diorders, Panic disorder, Agoraphobia, Social phobia, Generalized anxiety disorder, Simple phobia, Posttraumatic stress disorder
Diagnosis of stressor-related disorders assessed via CIDI Adjustment Disorder Module (Perkonigg et al., 2019) | Day 0, Month 6, Month 12
  Presence of Adjustment disorder is indicated with "yes" or "no" based on ICD-11 criteria.
Death anxiety assessed via Death and Dying Distress Scale (DADDS; Lo et al., 2011) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 6-point Likert scale from 0 (no distress) to 5 (extreme distress), with a total score ranging from 0 to 75. Higher scores indicate higher levels of death anxiety.
Dignity-related distress assessed via the Sense of Dignity Item (SDI; Chochinov et al., 2002) | Day 0, Month 3, Month 6, Month 9, Month 12
  Item is scord on a 7-point Likert-scale from 0 (no sense of loss of dignity) to 6 (extreme sense of loss of dignity).
Dignity-related distress assessed via the Patient Dignity Inventory (PDI; Chochinov et al., 2008) | Day 0, Month 3, Month 6, Month 9, Month 12
  The following subscales of the PDI are used: 1) Physical Symptom Distress, 2) Body Image and Loss of Autonomy. Items are scored on a 5-point Likert-scale from 0 (no problem) to 5 (an overwhelming problem). Higher scores indicate a higher sense of loss of dignity.
Quality of life assessed via the Quality of Life at the End of Life-Cancer-Psychosocial Questionnaire (QUAL-EC-P) | Day 0, Month 3, Month 6, Month 9, Month 12
  Subscales used: 1) Life completion, 2) Preparation for the end of life. Items are scored on a 5-point Likert scale from 0 (not at all) to 4 (completely), with a total score ranging from 0 to 36. Higher scores indicate higher quality of life.

OTHER OUTCOMES:
Prognostic awareness assessed via semistructured interview for subjective goal of oncological treatment (El-Jawahri et al., 2020; DeMartini et al., 2019) | Day 0, Month 6, Month 12
  Patients are asked about perceived goals of the cancer treatment and what they perceive to be their oncologists' goals for their treatment.
Subjective experience of end-of-life discussions with health care provider assessed via semi-structured interview (El-Jawahri et al., 2020) | Day 0, Month 3, Month 6, Month 9, Month 12
  Patients are asked whether they discussed their wishes regarding medical treatment with their oncologist and how they experienced these conversation.
Perceived relationship with healthcare provider assessed via Quality of Life at the End of Life-Cancer-Psychosocial Questionnaire (QUAL-EC-P) | Day 0, Month 3, Month 6, Month 9, Month 12
  Subscale Relationship with Healthcare Provider. Items are scored on a 5-point Likert scale from 0 (not at all) to 4 (completely), with a subscale score ranging from 0 to 20. Higher scores indicate a stronger relationship with health care providers.
Flexibility of coping with incurable cancer assessed via Loss Orientation and Life Engagement in Advanced Cancer Scale (LOLES; Vehling et al., 2018) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 5--point Likert scale from 0 (not at all) to 4 (nearly all the time). High scores indicate high levels of loss orientation, life engagement and coping efforts, respectively.
Receipt of medical treatment in last 30 days of life assessed via Medical Chart Review (Abedini et al., 2019) | Month 12
  Chemotherapy, immunotherapy, targeted therapy, hormonal therapy, inpatient treatment, emergency room visits, intensive care treatment, receipt of ambulatory or inpatient specialized or general palliative care
Subjective experience and psychological adaptation of family caregivers assessed via semistructured qualitative interviews, diagnostic interviews, and self-report questionnaires | Day 0, Month 3, Month 6, Month 9, Month 12
  Measures include a) identical versions of the measures used for patients, b) complementary versions of patient measures adapted for caregivers, c) caregiver-specific instruments
Desire for hastened death assessed via Schedule of Attitudes Toward Hastened Death (SAHD; Kolva et al., 2017) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored with either being true (1) or false (0). For the total score, number of endorsed items are counted, ranging from 0 to 6. Higher scores indicate higher levels of desire for hastened death.
Suicidality assessed via Beck Scale for Suicidal Ideation (BSS; Beck & Steer, 1993; Kliem & Brähler, 2015) | Day 0, Month 3, Month 6, Month 9, Month 12
  Intensity of suicidal tendencies is measured with three statements for each item. Statements are scored from 0 to 2. If screening items for active and passive suicidal ideation are scored with 0, participants are asked to skip to the items regarding previous suicidal attempts. The screening score ranges from 0 to 10, the total score ranges from 0 to 38. Higher values indicate stronger suicidal tendencies.
Depressive symptoms assessed via Patient Health Questionnaire-9 (PHQ-9; Kroenke et al., 2001) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 4--point Likert scale ranging from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 27. Scores ≥10 indicate moderate, scores ≥15 severe depression.
Anxiety symptoms assessed via Generalized Anxiety Disorder Questionnaire-7 (GAD-7; Spitzer et al., 2006) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 4--point Likert scale ranging from 0 (not at all) to 3 (nearly every day), with a total score ranging from 0 to 21. Scores ≥10 indicate moderate, scores ≥15 severe anxiety.
Adverse events assessed via Inventory for the Balanced Assessment of Negative Effects of Psychotherapy (INEP, Ladwig, Rief & Nestoriuc, 2014) | Month 3, Month 6, Month 9, Month 12, Weekly through treatment completion (median of 9 months)
  Six items are scored on a scale from 7-point scale from -3 (worsening) to 3 (improvement), fifteen items are scored on a 4-point Likert-scale from 0 (not at all) to 4 (completely). If patients attributed changes to the therapy itself, frequencies, means, and standard deviation of negative (-3 to 1), no (0), and positive changes (1 to 3) are calculated.
Adverse events assessed via therapy session protocols | Month 3, Month 6, Month 9, Month 12, Weekly through treatment completion (median of 9 months)
  Therapists document adverse events on a standardized form after each therapy session.
Therapeutic alliance assessed via Working Alliance Inventory - short revised (WAI-SR; Wilmers et al., 2024) | Month 3, Month 6, Month 9, Month 12, Weekly through treatment completion (median of 9 months)
  Items are scored on a 5-point Likert-scale from 1 (never) to 5 (always), with a total score ranging from 12 to 60. Higher scores indicate a stronger working alliance.
Agency assessed via Therapeutic Agency Inventory (TAI; Huber et al., 2019) | Weekly through treatment completion (median of 9 months)
  Items are scored on a 5-point Likert-scale from 1 (not true) to 5 (very true), with a total score ranging from 15 to 75. Higher scores indicate a stronger sense of agency.
Interpersonal problems assessed via Inventory of Interpersonal Problems - German Version (IIP-D-32; Horowitz et al., 1994) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 5-point Likert-scale from 0 (not) to 4 (very much), with the total score ranging from 0 to 128. Higher total scores indicate higher distress due to interpersonal problems.
Emotional dependence on others assessed via Depressive Experiences Questionnaire (DEQ; Blatt et al., 1976) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 7-point Likert scale from 1 (strongly disagree) to 7 (strongly agree), with a total score ranging from 18 to 126. Higher scores indicate higher dependence on others to regulate emotional distress.
Perceived communication in partnership assessed via Couple Communication Scale (CCS; Conrad et al., 2019) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree), with a total score ranging from 10 to 50. Higher scores indicate better communication in relationships.
Therapy adherence assessed via Penn Adherence/Competence Scale for Supportive-Expressive Dynamic Psychotherapy (Barber & Crits-Christoph, 1996), therapists' session protocols, supervision protocols, and therapists' diagnostic protocols | Weekly through treatment completion (median of 9 months)
  Rating by trained observers.
Insight into repetitive dysfunctional relationship patterns assessed via rating of therapy session transcripts with Insight into Conflictual Relationship Patterns Scale (ICR; Jennissen et al., 2020) | Weekly through treatment completion (median of 9 months)
  Trained observers rate each audio recorded therapy session on a 5-point Likert-scale from 0 (not at all) to 4 (very much), with a total score ranging from 0 to 48. Higher scores indicate a more complex understanding of internal states and interpersonal processes.
Defense mechanisms assessed via rating of therapy session transcripts with Defense Mechanisms Rating Scale (DMRS; Perry & Henry, 2004) | Weekly through treatment completion (median of 9 months)
  Therapy session transcripts are rated by trained observers, Items are scored on a 5-point Likert-scale from 0 (not at all) to 4 (very much). A percentage score of defensive functioning is calculated.
Perceived coping resources assessed via Questionnaire for Patient Competence in Coping with Cancer (PCQ, Aderhold et al., 2019) | Day 0, Month 3, Month 6, Month 9, Month 12
  Subscales used: 1) coping competence, 2) adaptability. Items are scored on a 6-point Likert scale from 0 (not at all) to 5 (completely), with a total score ranging from 0 to 35, and subscale scores ranging from 0 to 20 and 0 to 15. Higher scores indicate better coping.
Medical parameters of oncological disease and treatment | Day 0, month 6, month 12
  Day 0: Tumor site, date of first diagnosis, type of disease, date of diagnosis of recurrence/second tumor, stage of disease, Charlson Comorbidity Index (CCI); Day 0, month 6 and month 12: oncological treatments received, number of therapy lines, psychopharmacological medication, performance status (ECOG Status/Karnofsky Index), presence and date of disease progression
Physical symptom distress assessed via Memorial Symptom Assessment Scale - Short Form (MSAS-SF; Chang et al., 2000) | Day 0, Month 3, Month 6, Month 9, Month 12
  Items are scored on a 5-point Likert-scale ranging from 0 (not at all distressed) to 4 (very much distressed). The average symptom score is calculated. Higher scores indicate higher physical symptom burden.
Frequency and technique of psychooncological treatment assessed via semistructured interview and modified version of Multitheoretical List of Therapeutic Interventions-30 (Solomonov et al., 2019) | Day 0, Month 3, Month 6, Month 9, Month 12
  Scale expanded by frequent intervention techniques used in psycho-oncologyícal treatments. Items are scored on a 5-point Likert-scale from 1 (not at all typical of the session) to 5 (very typical of the session), with a total score ranging from 39 to 195. Higher scores indicate a rather typical use of intervention techniques.
Type and frequency of utilization of other psychosocial support services assessed via semistructured interview | Day 0, Month 6, Month 12

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Clinical Institute for Psychosomatic Medicine and Psychotherapy, University Medical Center Düsseldorf, Düsseldorf
  - University Medical Center Hamburg-Eppendorf, Hamburg
  - Psychosomatics, Psychotherapy and Psychooncology, Medicine II, University of Würzburg, Würzburg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Philipp R, Walbaum C, Lindner R, Karger A, Maatouk I, Dinger U, Vehling S. [ORPHYS - Treatment Manual for a Short-Term Psychodynamic Psychotherapy in Patients with Serious Physical Illness]. Psychother Psychosom Med Psychol. 2024 Aug;74(8):345-351. doi: 10.1055/a-2322-8596. Epub 2024 Jun 17. German. PMID 38885656
- [Background] Perkonigg A, Strehle J, Beesdo-Baum K, Lorenz L, Hoyer J, Venz J, Maercker A. Reliability and Validity of a German Standardized Diagnostic Interview Module for ICD-11 Adjustment Disorder. J Trauma Stress. 2021 Apr;34(2):275-286. doi: 10.1002/jts.22597. Epub 2020 Nov 5. PMID 33151596
- [Background] Huber J, Nikendei C, Ehrenthal JC, Schauenburg H, Mander J, Dinger U. Therapeutic Agency Inventory: Development and psychometric validation of a patient self-report. Psychother Res. 2019 Oct;29(7):919-934. doi: 10.1080/10503307.2018.1447707. Epub 2018 Mar 20. PMID 29557306
- [Background] Brahler E, Horowitz LM, Kordy H, Schumacher J, Strauss B. [Validation of the Inventory for Interpersonal Problems (IIP). Results of a representative study in East and West Germany]. Psychother Psychosom Med Psychol. 1999 Nov;49(11):422-31. German. PMID 10593141
- [Background] Galushko M, Strupp J, Walisko-Waniek J, Hahn M, Loffert S, Ernstmann N, Pfaff H, Radbruch L, Nauck F, Ostgathe C, Voltz R. Validation of the German version of the Schedule of Attitudes Toward Hastened Death (SAHD-D) with patients in palliative care. Palliat Support Care. 2015 Jun;13(3):713-23. doi: 10.1017/S1478951514000492. Epub 2014 May 22. PMID 24849188
- [Background] El-Jawahri A, Forst D, Fenech A, Brenner KO, Jankowski AL, Waldman L, Sereno I, Nipp R, Greer JA, Traeger L, Jackson V, Temel J. Relationship Between Perceptions of Treatment Goals and Psychological Distress in Patients With Advanced Cancer. J Natl Compr Canc Netw. 2020 Jul;18(7):849-855. doi: 10.6004/jnccn.2019.7525. PMID 32634779
- [Background] Conrad M, Engelmann D, Friedrich M, Scheffold K, Philipp R, Schulz-Kindermann F, Harter M, Mehnert A, Koranyi S. [Assessment of Couples' Communication in Patients with Advanced Cancer: Validation of a German Version of the Couple Communication Scale (CCS)]. Psychother Psychosom Med Psychol. 2019 May;69(5):189-196. doi: 10.1055/a-0583-4837. Epub 2018 Apr 13. German. PMID 29653458
- [Background] Hack TF, McClement SE, Chochinov HM, Cann BJ, Hassard TH, Kristjanson LJ, Harlos M. Learning from dying patients during their final days: life reflections gleaned from dignity therapy. Palliat Med. 2010 Oct;24(7):715-23. doi: 10.1177/0269216310373164. Epub 2010 Jul 6. PMID 20605851
- [Background] Abedini NC, Hechtman RK, Singh AD, Khateeb R, Mann J, Townsend W, Chopra V. Interventions to reduce aggressive care at end of life among patients with cancer: a systematic review. Lancet Oncol. 2019 Nov;20(11):e627-e636. doi: 10.1016/S1470-2045(19)30496-6. PMID 31674321
- [Background] Vehling S, Gerstorf D, Schulz-Kindermann F, Oechsle K, Philipp R, Scheffold K, Harter M, Mehnert A, Lo C. The daily dynamics of loss orientation and life engagement in advanced cancer: A pilot study to characterise patterns of adaptation at the end of life. Eur J Cancer Care (Engl). 2018 Jul;27(4):e12842. doi: 10.1111/ecc.12842. Epub 2018 Apr 27. PMID 29700876
- [Background] Koranyi S, Hinz A, Hufeld JM, Hartung TJ, Quintero Garzon L, Fendel U, Letsch A, Rose M, Esser P, Mehnert-Theuerkauf A. Psychometric Evaluation of the German Version of the Demoralization Scale-II and the Association Between Demoralization, Sociodemographic, Disease- and Treatment-Related Factors in Patients With Cancer. Front Psychol. 2021 Nov 24;12:789793. doi: 10.3389/fpsyg.2021.789793. eCollection 2021. PMID 34899543